CLINICAL TRIAL: NCT04495244
Title: Investigation of a Novel Blood Test to Identify Breast Cancer (IDBC)
Brief Title: A Study to Identify Breast Cancer (IDBC)
Acronym: IDBC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Syantra Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 241391
Record Dates: First submitted 2020-07-07; First posted 2020-07-31 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Breast Cancer Female
Keywords: Detection, blood test, clinical assay

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — Whole blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Investigational Population: Suspected Invasive Breast Cancer (any size) or DCIS (pre-invasive) are of particular interest. Women with abnormal screening mammograms (R3-5) recalled for further investigation.
  Inclusion criteria
  * Women with suspected Invasive Breast Cancer (tumours of any size and/or DCIS).
  * Individuals with an abnormal or suspicious screening mammogram recalled for further evaluation.
  * Suspected Invasive Breast Cancer (tumours of any size and/or DCIS).
  * Willing to give written Informed Consent and provide whole blood samples
  * Age 30-75 years
  Exclusion criteria
  * Breast surgery within the previous 12 months (for any reason) or recent breast biopsy (including needle core biopsy)
  * Inoperable (T4 category) or inflammatory breast cancer
  * Previous history of cancer previously at any site
  * Previous history of breast cancer
  * Concomitant or other concurrent anti-cancer therapy
  * Male
  * No histopathological diagnosis
  Interventions: Diagnostic Test: Syantra DX Breast Cancer
- Borderline (Atypica and LCIS) Population: Women with borderline pathological B3 lesions (suspected atypia Ductal or Lobular and benign proliferative disease without DCIS or invasion) Inclusion criteria
  * Abnormal screening mammogram with suspected benign breast disease or proliferative changes
  * Willing to give Written Informed Consent and provide whole blood samples
  * Aged 30-75 years
  Exclusion criteria
  * Existing cancer diagnosis
  * Male
  * Breast surgery within the previous 12 months (for any reason) or recent breast biopsy (including needle core biopsy)
  * Previous history of any cancer
  * Previous history of breast cancer
  * Concomitant or other concurrent anti-cancer therapy
  Interventions: Diagnostic Test: Syantra DX Breast Cancer
- Control Population: Healthy Controls Inclusion criteria
  * Normal breast examination - No cancer detected/suspected by physical exam, diagnostic radiology or screening mammography
  * Willing to give Written Informed Consent and provide whole blood samples
  * Aged 30-75 years
  Exclusion criteria
  * Cancer diagnosis
  * Male
  * Breast surgery within the previous 12 months (for any reason) or recent breast biopsy (including needle core biopsy)
  * Previous history of any cancer
  * Concomitant or other concurrent anti-cancer therapy
  Interventions: Diagnostic Test: Syantra DX Breast Cancer

INTERVENTIONS:
Diagnostic Test: Syantra DX Breast Cancer — Blood test for detecting the presence of breast cancer.

SUMMARY:
Detecting cancer as early as possible is key to achieving positive outcomes in response to diagnosis and treatment. The current project is aimed at validating a novel blood-based breast cancer identification test (Syantra DX Breast Cancer) that has been developed by Syantra Inc. Syantra DX Breast Cancer measures gene expression signatures in whole blood, and has been retrospectively demonstrated in 780 samples. The test uses proprietary algorithms to analyse gene expression characteristics from a novel multi-biomarker panel, and then classify a sample as positive or negative for breast cancer. Based upon test performance in a retrospective environment, a prospective validation study is being proposed.

The primary objective of this study is to validate Syantra DX Breast Cancer methodology and biomarker panel using prospective samples, well categorized by diagnostic imaging scores, pathology outcomes, and subject characteristics.

DETAILED DESCRIPTION:
The current project is aimed at validating Syantra DX Breast Cancer in a UK population. Results of the UK study will be combined with those from additional sites, including those in Canada, with additional samples expected from the United States and South Korea. Syantra DX Breast Cancer measures gene expression signatures in whole blood, and has been retrospectively demonstrated in 780 samples. The test uses proprietary algorithms to analyse gene expression characteristics from a novel multi-biomarker panel, and then classify a sample as positive or negative for breast cancer. Based upon test performance in a retrospective environment, a prospective validation study is being proposed, and is described below.

The study seeks to evaluate performance of Syantra DX Breast Cancer in prospective samples and to optimize test methodology and biomarkers. Key to performance of the study is recruitment of women who have received an abnormal mammography report, and have been classified under the UK Royal College of Radiologists Breast Group (RCRBG) scoring system in categories 3 - 5. This will support the ability to employ the test for breast cancer detection in a screening/call-back environment. To complete the study cohort, additional women will be recruited from the population who have normal or benign mammography results (RCRBG category 1 and 2), and/or a recent normal physical breast exam, with no history of breast cancer. Blood samples will be acquired from all women following completion of an informed consent procedure.

For those with an abnormal mammogram, blood will be drawn before a biopsy is performed. All sample information will be de-identified, and the samples will be processed and analysed according to Syantra DX Breast Cancer standard operating procedures. These procedures include extracting sample RNA and aliquoting for storage in a manner that maintains sample anonymity. All processing and analysis will be conducted in a blind environment without knowing the associated RCRBG or pathology outcomes for any samples. Only after testing is complete will sample classifications be revealed. Syantra DX Breast Cancer results will then be compared to RCRBG, biopsy and pathology data to determine concordance, and statistics will be calculated. If or when biomarker panel or test methodology is modified during the performance of the study, samples will be reanalysed with updated test parameters. This reanalysis will make use of a de-identified aliquot of sample RNA to ensure that testing is maintained in a blind environment.

There is an optional part of the study procedure that is included as 'additional research'. A specific question seeking approval for the additional research is included on the study consent form. For individuals who agree to participate in the additional research, material extracted from their blood sample will be stored for additional investigations.

ELIGIBILITY:
Inclusion criteria

* Aged 30-75 years
* Normal breast examination - No cancer detected/suspected by physical exam, diagnostic radiology or screening mammography
* Women with suspected Invasive Breast Cancer
* Individuals with an abnormal or suspicious mammogram
* Abnormal screening mammogram with suspected benign breast disease or proliferative changes

Exclusion criteria

* Cancer diagnosis
* Male
* Breast surgery within the previous 12 months (for any reason) or recent breast biopsy (including needle core biopsy)
* Previous history of any cancer
* Concomitant or other concurrent anti-cancer therapy
* Inoperable or inflammatory breast cancer

Ages: 30 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-identified
Study Population: Populations will be selected from women visiting the Nightingale Centre at Wythenshaw Hospital for breast cancer imaging.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2019-01-24 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Performance of the Syantra DX Breast Cancer test as assessed by sensitivity and specificity | through completion of the study, approximately eighteen months
  The number of participants that test positive or negative for breast cancer with the Syantra DX Breast Cancer test and their breast cancer status as assessed by mammography or pathology.

SECONDARY OUTCOMES:
Modulate test methodology to account for differences between retrospective and prospective samples | through completion of the study, approximately eighteen months
  Determine the sensitivity and specificity of the assay with biomarker panel modifications.
Performance of the Syantra DX Breast Cancer test in prediction of molecular subtype of breast cancer as assessed by pathology | through completion of the study, approximately eighteen months
  Correlate the performance of the test to molecular characterizations of identified cancers as assessed by pathology of tissue from biopsy or resection.

CONTACTS AND LOCATIONS:
Overall Officials: Nigel Bundred, MD, Principal Investigator — Manchester University NHS Foundation Trust; Cliona Kirwin, MD, Study Director — Manchester University NHS Foundation Trust
Locations (1):
- Wythenshawe Hospital, Southmoor Road, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No